CLINICAL TRIAL: NCT06050369
Title: Actimetric and Electrophysiological Analyses of Repetitive Behaviors (Tics and Compulsions)
Brief Title: Objective Characterizatoion of Repetitive Behaviors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C21-48; 2022-A01332-41 (Registry Identifier: ID RCB)
Record Dates: First submitted 2023-04-28; First posted 2023-09-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: OCD; Tic Disorders; Gilles de la Tourette Syndrome
Keywords: Electrophysiology; Electroencephalogram; EEG; Accelerometer; Biomarker; Symptom provocation
MeSH Terms: conditions — Tic Disorders; Tourette Syndrome | interventions — Electroencephalography; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GTS group (Experimental): This arm will be studied to get some electrophysiological marker of tics. The patients will be their own control (periods with symptoms vs. free symptoms periods).
  Interventions: Device: EEG; Device: MRI
- OCD group (Experimental): This arm will be studied to get some electrophysiological marker of compulsions. The patients will be their own control (periods with symptoms vs. free symptoms periods).
  Interventions: Device: EEG; Device: MRI

INTERVENTIONS:
Device: EEG — Recording, from the scalp, the electrophysiological activity of the brain.
  Other Names: Electroencephalogram
Device: MRI — Get the anatomical shape of the brain.
  Other Names: magnetic resonance imaging

SUMMARY:
Introduction:

Repetitive behaviors (RB) constitute a broad range of symptoms across different psychiatric/neurologic disorders. The most famous are stereotypies (found in autism), compulsions (found in obsessive-compulsive-disorder, OCD) and tics (found in Gilles de la Tourette syndrome, GTS). For some patients, it is sometime difficult to distinguish the nature of the repetitive behaviors presented, however this distinction is crucial in order to chose the appropriate treatment.

Aim:

In our study, the investigators will try to define electrophysiological and accelerometric marker of both OCD and tics to allow objective distinction between both tics and compulsions.

Method:

Subjects: Both OCD and GTS patients will be recruited, 25 patients in each group.

Protocol: our study protocol will involve two step: a step in laboratory, another step at patient home.

* first step: both patients group will be recorded through a high density EEG and a portative EEG while doing a task of symptom provocation. Then they will get an anatomical MRI for source recontruction. Finally, the patients will have to mimic their symptom while wearing an accelerometer (a smartwatch).
* second step: both patient groups will be recorded at home through a portative EEG while tagging their symptom through a smartwatch (also used for accelerometry). After the recording, the patients will keep the smartwatch for 2 weeks, still tagging their sympoms (compulsions or tics).

ELIGIBILITY:
Inclusion Criteria:

* To be more of 15 years old or less than 65 years old
* To suffer from OCD and/or GTS (depressive, anxious and attention deficit hyperactivity disorder (ADHD) comorbidities are accepted)
* To be registered to the french social security (or something equivalent)
* To give written consent to participate to the research
* To have contraception for women participants (or to not have any sexual activity)

Exclusion Criteria:

* Patients with any other psychiatric disorders than those mentioned in the inclusion criteria
* Patients with any other neurological disorder than GTS
* Patients who are not able to take decisions for themselves
* Pregnant women
* Patients not allowed to get MRI due to contraindication
* Patients not speaking french

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-28 (Actual); Primary Completion 2027-12-27 (Estimated); Study Completion 2027-12-27 (Estimated)

PRIMARY OUTCOMES:
modification of power (μV2) in EEG frequencies before compulsions in Obsessive-Compulsive Disorder patients | one year
  change in the power EEG frequencies in OCD patients before compulsions EEG frequencies come to 0 to 250 Hz, the power is the amplitude of oscillations
modification of power (μV2) in EEG frequencies before tics in Gilles de la Tourette patients | one year
  change in the power of EEG frequencies in GTS patients before tics EEG frequencies come to 0 to 250 Hz, the power is the amplitude of oscillations

SECONDARY OUTCOMES:
Difference in power (μV2) in EEG frequencies between obsessive-compulsive disorder patients and Gilles de la Tourette patients | One year and a half
  Difference in the power in the EEG frequencies between obsessive-compulsive disorder patients and Gilles de la Tourette patients EEG frequencies come to 0 to 250 Hz, the power is the amplitude of oscillations
percentage (%) of compulsions and tics detected by accelerometer | One year and a half
  percentage of compulsions and tics detected by accelerometer
Correlation of EEG frequency power (arbitrary units) detected before compulsions and scores get with clinical scales (Y-BOCS) | One year and a half
  Correlation between power in EEG frequencies and Y-BOCS score get by each individual patients Y-BOCS = Yale-Brown Obsessive-Compulsive Scale; Scores range from 0 to 40 with 40 corresponding to the maximum severity of symptoms
Correlation between number of compulsions detected by accelerometer and Y-BOCS scores get by obsessive-compulsive patients | One year and a half
  Correlation between number of compulsions detected by accelerometer and Y-BOCS scores get by obsessive-compulsive patients Y-BOCS = Yale-Brown Obsessive-Compulsive Scale; Scores range from 0 to 40 with 40 corresponding to the maximum severity of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Luc MALLET, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - Hôpital Albert Chenevier, Créteil
  - Hôpital Henri Mondor, Créteil
  - Hôpital Pitié Salpêtrière, Paris